CLINICAL TRIAL: NCT07007364
Title: Neoadjuvant Low-Dose Radiotherapy Combined With Adebrelimab and Single-Agent Albumin-Bound Paclitaxel Chemotherapy for Early-Stage Oral Squamous Cell Carcinoma: A Prospective, Single-Arm Clinical Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jun Jia (Other)
Responsible Party: Sponsor-Investigator, Jun Jia, Director, Hospital of Stomatology, Wuhan University
Organization: Hospital of Stomatology, Wuhan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HStomatologyWuhan2
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Early-Stage Oral Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant low-dose radiotherapy combined with adebrelimab and monotherapy with albumin paclitaxel (Experimental): Eligible patients received neoadjuvant low-dose radiotherapy combined with Adebrelimab and monotherapy with albumin paclitaxel for two cycles. Radical surgical resection is planned to be carried out 3 to 4 weeks after neoadjuvant therapy. Patients who obtain PCR after evaluation by the researchers after the operation will be maintained for 6 cycles of immunomonotherapy
  Interventions: Drug: Adebrelimab Combined With Albumin Paclitaxel

INTERVENTIONS:
Drug: Adebrelimab Combined With Albumin Paclitaxel — Eligible patients received neoadjuvant low-dose radiotherapy combined with Adebrelimab and monotherapy with albumin paclitaxel for two cycles. Radical surgical resection is planned to be carried out 3 to 4 weeks after neoadjuvant therapy. Patients who obtain PCR after evaluation by the researchers after the operation will be maintained for 6 cycles of immunomonotherapy

SUMMARY:
This is a prospective, single-arm, Phase II clinical trial. The included population consisted of untreated patients with histologically confirmed stage I-II oral squamous cell carcinoma. Eligible patients received neoadjuvant low-dose radiotherapy combined with adibelizumab and monotherapy with albumin paclitaxel for two cycles. Radical surgical resection is planned to be carried out 3 to 4 weeks after neoadjuvant therapy. Patients who obtain PCR after evaluation by the researchers after the operation will be maintained for 6 cycles of immunomonotherapy. The primary endpoints were the rate of pathological response and the rate of exemption from cervical lymph node dissection. The secondary endpoints included progression-free survival, local control rate, distant metastasis-free rate, overall survival, safety and quality of life of patients, as well as the exploration of biomarkers

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 70, gender not limited;
2. Confirmed by pathological examination as oral squamous cell carcinoma (anterior 2/3 of the tongue, floor of the mouth, gingiva, buccal mucosa, hard palate, posterior molar area);
3. Diagnosed as stage I-II oral squamous cell carcinoma (T1-2N0M0) according to the 8th edition of the clinical staging system of the American Joint Committee on Cancer;
4. ECOG 0-1 point;
5. Vital organs function normally and can tolerate the prescribed treatment plan:

   1. There was no obvious abnormality in bone marrow hematopoietic function before treatment: white blood cell count ≥3.5×109/L, neutrophil count ≥2.0×109/L; Hemoglobin ≥100g/L Platelet count ≥100×109/L;
   2. No obvious abnormalities were observed in liver and kidney functions before treatment: Total bilirubin ≤1.5 times the upper limit of normal; Aspartate aminotransferase and/or alanine aminotransferase ≤2.5 times the normal upper limit; Alkaline phosphatase ≤2.5 times the normal upper limit; Creatinine clearance rate ≥60 mL/min;
   3. The examination results of thyroid function, coagulation function, pituitary function, inflammatory infection indicators, myocardial enzymes, electrocardiogram and echocardiography are normal;
6. Women of childbearing age (18-49 years old) have negative serum or urine HCG tests within 7 days before treatment and agree to use medically approved contraceptive measures during the treatment period and within 120 days after the end of treatment;
7. Sign the informed consent form, voluntarily participate in the clinical trial research project, and be willing and able to comply with the follow-up, treatment, laboratory testing and other research requirements stipulated in the research schedule.

Exclusion Criteria:

* 1. There is uncontrollable pleural effusion, pericardial effusion or peritoneal effusion that requires repeated drainage; 2. There is a history of allergy to adbelimab in the past; 3. Has received any of the following treatments:

  1. Having received any other investigational drugs within 4 weeks before the first use of the investigational drug or no more than 5 half-lives from the last investigational drug use;
  2. Enroll in another clinical study simultaneously, unless it is an observational (non-interventional) clinical study or follow-up of an interventional clinical study;
  3. Have received anti-tumor treatment (including radiotherapy, chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biological therapy or tumor embolization) within 2 weeks before the first use of the study drug;
  4. Subjects who need to be given corticosteroids (an equivalent dose of > 10 mg prednisone per day) within 2 weeks before the first use of the study drug. Hormones are allowed for routine chemotherapy pretreatment without the need to adjust the dosage. In other special circumstances, communication with the researcher is required. In the absence of active autoimmune diseases, inhaled or topical use of steroids and adrenal cortical hormones with a dose of ≤10 mg/ day of prednisone as an therapeutic dose is permitted.
  5. Those who have received anti-tumor vaccines or those who have received live vaccines within 4 weeks before the first administration of the study drug;
  6. Underwent major surgery or suffered severe trauma within 4 weeks before the first use of the study drug;
  7. Patients who have previously received treatment with taxanes; 4. The toxicity of previous anti-tumor treatments has not recovered to ≤CTCAE 5.0 grade 1 (except for alopecia) or the level specified in the inclusion/exclusion criteria; 5. Have active autoimmune diseases or a history of autoimmune diseases (such as interstitial pneumonia, colitis, liver inflammation, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to the above diseases or syndromes); Excluding patients with vitiligo or childhood asthma/allergies that have been cured and do not require any intervention in adulthood; Autoimmune hypothyroidism treated with a stable dose of thyroid replacement hormone; Type 1 diabetes using a stable dose of insulin; 6. Have a history of immunodeficiency, including a positive HIV test, or having other acquired or congenital immunodeficiency diseases, or having a history of organ transplantation and allogeneic bone marrow transplantation, or active hepatitis (hepatitis B reference: HBV DNA test value exceeds 500 IU/ml or 2500 copies /mL); 7. The subjects have poorly controlled cardiovascular clinical symptoms or diseases, including but not limited to: such as: (1) NYHA grade II or above heart failure; (2) Unstable angina pectoris (3) Had a myocardial infarction within one year; (4) Supraventricular or ventricular arrhythmias of clinical significance that have not undergone clinical intervention or remain poorly controlled after clinical intervention; 8. Severe infections (CTCAE 5.0 > 2) occurred within 4 weeks before the first use of the study drug, such as severe pneumonia requiring hospitalization, bacteremia, and complications of infection, etc. Baseline chest imaging examinations indicated the presence of active pulmonary inflammation, symptoms and signs of infection within 2 weeks before the first use of the study drug, or the need for oral or intravenous antibiotic treatment, excluding the cases of preventive antibiotic use.

     9. Have a history of interstitial lung disease (except for radiation pneumonitis and non-infectious pneumonia that have not received hormone therapy); 10. Patients who were found to have active pulmonary tuberculosis infection through medical history or CT examination, or those who had a history of active pulmonary tuberculosis infection within one year before enrollment, or those who had a history of active pulmonary tuberculosis infection more than one year ago but have not received formal treatment; 11. Any other malignant tumor was diagnosed within 5 years prior to the first use of the study drug, except for malignant tumors with a low risk of metastasis and death (5-year survival rate > 90%), such as adequately treated basal cell or squamous cell skin cancer or cervical carcinoma in situ; 12. Pregnant or lactating women; 13. As judged by the researcher, the subjects have other factors that may cause them to be forced to terminate the study halfway, such as suffering from other serious diseases (including mental disorders) requiring combined treatment, having severely abnormal laboratory test values, family or social factors that may affect the safety of the subjects or the collection of experimental data

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-19 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
MPR | From enrollment to the end of surgery,assessed up to 6 months
  The percentage of viable tumor cells remaining in the tumor bed after neoadjuvant therapy is ≤10%, regardless of whether viable tumor cells remain in the lymph nodes
The rate of exemption from cervical lymph node dissection surgery | From enrollment to the end of surgery,assessed up to 6 months
  During the operation, multiple biopsies were performed on the primary lesion. If no tumor cells were found, cervical lymph node dissection was waived

SECONDARY OUTCOMES:
PFS | From enrollment to the first appearance of disease progression or date of deathfrom any cause,whichever came first, assessed up to 36 months
  The calculation starts from the day of enrollment until treatment failure, death due to any cause, or the last follow-up occurs, with the first occurrence as the endpoint
LRFS | From enrollment to the first appearance of disease progression or date of deathfrom any cause,whichever came first, assessed up to 36 months
  The calculation starts from the day of enrollment until local and/or regional recurrence occurs or at the last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Stomatology, Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No